CLINICAL TRIAL: NCT01626053
Title: The Efficacy and Treatment Adherence With an Integrated Program on HbA1c Scores in Patients With Type 2 Diabetes
Acronym: ASMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KRJG Services Inc. (Other)
Collaborators: K21 Health Foundation (Other); Kosciusko County Health Department (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ASMART-01; 2008-4-03 (Other Grant/Funding Number: K21 Health Foundation)
Record Dates: First submitted 2012-06-07; First posted 2012-06-22 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: psychological; intervention; stages of change; motivational interviewing; coping skills; HbA1C; psychological testing; integrated care; behavioral health
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention)
  Interventions: Other: Control Group
- lifestyle counseling (Experimental): These participant received the ASMART interventions.
  Interventions: Behavioral: ASMART

INTERVENTIONS:
Behavioral: ASMART — Motivational Interviewing, Stages of Change, Psychological Testing, Bio-psychosocial assessment, responsive diabetes education, support, Cognitive-behavioral interventions
  Arms: lifestyle counseling
Other: Control Group — no intervention
  Arms: control group

SUMMARY:
It is hypothesized for this study that the coupling of the Millon Behavioral Medicine Diagnostic, biopsychosocial evaluation, motivational interviewing, relapse prevention, and ongoing support can produce improved outcomes with diabetics who have previously been unsuccessful with the traditional care. This study examined the relationship between patients' HbA1c levels and patients' involvement in the ASMART program, a multifaceted program involving psychological intervention. The study was conducted through the Kosciusko Health Department and funded by K21 Health Foundation.

DETAILED DESCRIPTION:
The study involved 182 Type 2 Diabetes patients with an HbA1c score above 7, reflecting poor control of diabetes. The experimental group consisted of 124 patients who joined the ASMART program, while the control group consisted of 60 patients who continued to receive traditional care. Statistical analysis involved comparing pretest & posttest HbA1c levels for the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes patients with an HbA1c score over 7

Exclusion Criteria:

* No Type 1 patients
* No children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes in A1c levels for pretest and post test (Preset baseline and post-test 2 years | Pretest / posttest
  Statistical analysis involved comparing pretest and psttest HbA1c levels for the experimental group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Kevin W Roberts, PsyD, Principal Investigator — Grace College; Dana L Coates, D.O., Study Director — Kosciusko Community Hospital
Locations (1):
- Northern Lakes Medicine, Warsaw, Indiana, United States